CLINICAL TRIAL: NCT03723473
Title: Peripheral Artery Disease: Gated P-31 Magnetic Resonance Spectroscopy in Functional Assessment of Peripheral Artery Disease (spectroAMI)
Brief Title: Spectroscopy in Functional Assessment of Peripheral Artery Disease (spectroAMI)
Acronym: SPECTROAOMI
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Dr MAYER Ronald A. Department of Physiology, Michigan State University (Unknown); Dr SLADE Jill M. Department of Osteopathic Manipulative Medicine, Michigan State University (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1708029; 2017-A01421-52 (Other: ANSM)
Record Dates: First submitted 2018-10-26; First posted 2018-10-29 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Arterial Occlusive Diseases
Keywords: Peripheral Arterial Occlusive Disease (PAOD); Phosphorus-31; Magnetic Resonance Imaging (MRI); Spectroscopy; Revascularization; Claudication with surgical planning
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Arterial Occlusive Disease 1 | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAOD patients statin (+): Patients with Peripheral Arterial Occlusive Disease (PAOD) and statin treatment.
  They will have Magnetic Resonance Imaging (MRI; muscular volume and composition) and gated-P-31 magnetic resonance spectroscopy (MRS) with low-intensity ergometric exercise. It will be performed before surgery (within 48h) and after surgery (first week)
  Interventions: Device: Magnetic Resonance Imaging (MRI)
- PAOD patients statin (-): Patients with Peripheral Arterial Occlusive Disease (PAOD) without statin treatment .
  They will have Magnetic Resonance Imaging (MRI ; muscular volume and composition) and gated-P-31 magnetic resonance spectroscopy (MRS) with low-intensity ergometric exercise. It will be performed before surgery (within 48h) and after surgery (first week)
  Interventions: Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) — MRI (muscular volume and composition) and gated-P-31 magnetic resonance spectroscopy (MRS) with low-intensity ergometric exercise.

SUMMARY:
To explore the reliability of P-31 MR spectroscopy mitochondrial function in patients with peripheral arterial occlusive disease.

DETAILED DESCRIPTION:
Peripheral arterial occlusive disease (PAOD) is defined as the partial or total obstruction of one or more lower extremity arteries, most often of atherosclerotic origin. It is a common disease whose 5-years mortality is near 30%.The positive diagnosis is based on clinical examination and measurement of the ankle-brachial index (ABI), which is the ratio of systolic pressure of ankle and brachial systolic pressure. The threshold value for the diagnosis is <0.90. Physiopathologically, mitochondria have the predominant role of providing the ATP necessary for the energetic needs of myocytes, which increase drastically during muscle contraction during exercise. This energy production is of course conditioned by the availability of oxygen. In patients with PAOD, the decrease in blood flow secondary to significant stenosis has the direct consequence of disrupting oxygen delivery to distal muscles and thus limiting muscular performance. Because mitochondrial respiration is the only metabolic pathway capable of providing the energy needed to sustain an effort of several minutes, intermittent claudication in PAOD has logically been related to a hemodynamic mechanism of intermittent muscle hypoperfusion. Recently, an increasing number of histological or functional studies have suggested that episodes of ischemia-reperfusion could induce mitochondrial dysfunction. Medical treatment of patients frequently includes statins while a direct deleterious effect on mitochondrial function has been suspected, inducing a deterioration of the muscular oxidative capacity which would increase the factors hemodynamics and may accumulate in mitochondrial myopathy. In the light of these elements, it is clear that there would be a benefit in being able to distinguish and quantify 1) the part of the reduction of mitochondrial activity secondary to the hemodynamic factor alone due to a decreased muscle perfusion 2) the mitochondrial involvement (mitochondriopathy) potentially induced by oxidative stress in PAOD. 2 sub-groups are distinguished to identify the statin-induced mitochondrial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral arterial occlusive disease (PAOD) with claudication and surgery planning with proximal lesion (iliac or femoral (x-ray angiography or CT or MRA) and no distal lesions (doppler)
* ABI<0.90 or >1.30
* signed consent form
* health insurance coverage

Exclusion Criteria:

* Contraindication in the practice of MRI: pacemaker, metallic cardiac valve, intra-ocular metal part, claustrophobia
* critical ischemia >15 days
* Type 1 or 2 diabetes
* weight >200kg
* non stabilized hypertension
* beta-blockers
* non-atherosclerotic vascular occlusive disease (Buerger disease, Takayasu disease, venous disease, trapped popliteal artery etc..)
* Neurological pathology/non-voluntary contraction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Peripheral arterial occlusive disease with claudication and surgery planning
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Muscle phosphocreatine (PCr) recovery time constant | During the MRI procedure
  Muscle phosphocreatine (PCr) recovery time constant (index of muscle aerobic capacity) after gated low-intensity exercise (2"maximum voluntary isometric dorsiflexion contractions, at 30s intervals for 8min (total contractions = 15)

SECONDARY OUTCOMES:
Muscular volume and content | During the MRI procedure
  impact of muscular volume and content. Measures will be extracted from DIXON and T2* MRI
PCr recovery time constant | During the MRI procedure
  impact of statin treatment on PCr recovery time constant

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CROISILLE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No